CLINICAL TRIAL: NCT06731738
Title: A Phase 2 Proof-of-Concept Clinical Trial to Quantify Myocardial Manganese Uptake Rate by Cardiovascular Magnetic Resonance Imaging Following Mangafodipir Trisodium Administration in Healthy Volunteers and Heart Failure Patients With Preserved Ejection Fraction Caused by Hypertrophic Cardiomyopathy or Cardiac Amyloidosis.
Brief Title: Mangafodipir - an Intracellular Contrast Agent for Magnetic Resonance Imaging (MRI): Measuring Manganese Uptake Rate in Heart Failure Patients With Preserved Ejection Fraction (HFpEF) Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IC TARGETS AS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MNC001; 2023-508118-40-01 (EU CTIS Number)
Record Dates: First submitted 2024-11-25; First posted 2024-12-12 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFPEF)
Keywords: Mangafodipir; HFpEF; CMR; Heart Failure; Heart Disease; Manganese-enhanced magnetic resonance imaging (MEMRI)
MeSH Terms: conditions — Heart Failure; Heart Diseases | interventions — N,N'-bis(pyridoxal-5-phosphate)ethylenediamine-N,N'-diacetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HFpEF with HCM (Experimental): Heart failure patients with preserved ejection fraction caused by hypertrophic cardiomyopathy.
  Participants will have 2 cardiac MRIs (gadolinium- and manganese-enhanced) at Visit 2 and Vist 3, respectively.
  Interventions: Drug: Gadoteric acid; Drug: Mangafodipir trisodium injection
- HFpEF with CA (Experimental): Heart failure patients with preserved ejection fraction caused by cardiac amyloidosis.
  Participants will have 2 cardiac MRIs (gadolinium- and manganese-enhanced) at Visit 2 and Vist 3, respectively.
  Interventions: Drug: Gadoteric acid; Drug: Mangafodipir trisodium injection
- Healthy Volunteers (Experimental): Participants will have 2 cardiac MRIs (gadolinium- and manganese-enhanced) at Visit 2 and Vist 3, respectively.
  Interventions: Drug: Gadoteric acid; Drug: Mangafodipir trisodium injection

INTERVENTIONS:
Drug: Gadoteric acid — A gadolinium-based contrast agent (authorised auxiliary medicinal product (AMP)) will be injected i.v. at a dose of 0.2 mmol Gd/kg bw and T1 mapping and ECV measurement will be done.
Drug: Mangafodipir trisodium injection — Mangafodipir trisodium injection (IMP) will be administered i.v. at a dose of 5 µmol/kg bw and T1 mapping, Saturation Recovery T1 weighted imaging for measurement of the uptake rate, and T2 mapping, will be done.

SUMMARY:
More than half of heart failure patients have preserved ejection fraction (HFpEF), a condition caused by increased wall stiffness that impairs proper heart filling. Two types of cardiac fibrosis, replacement fibrosis and interstitial fibrosis, contribute to this stiffening. In addition, altered calcium handling in the cardiomyocytes is relevant. The currently available contrast agents in Magnetic Resonace Imaging (MRI) primarily detect cell loss caused by replacement fibrosis, and measurements of the extracellular volume provide clues about the status of interstitial fibrosis. However, the planned trial aims to utilise mangafodipir trisodium to measure cellular function independent of the impact of fibrosis. This information could be vital for accurate diagnosis, selection and monitoring of therapy. In addition, manganese-enhanced magnetic resonance imaging (MEMRI) may be used as an alternative to examinations with gadolinium-based contrast agents in the future.

DETAILED DESCRIPTION:
The trial is an open-label, single centre, Phase 2A, Proof-of-Concept (PoC) trial in adult male and female patients without randomisation.

Overall, up to 42 participants will be enrolled in this trial:

* A run-in phase will include up to 6 participants (healthy volunteers and HFpEF patients regardless of aetiology (HCM, CA).
* The main phase of the trial will include 12 HFpEF with HCM, 12 HFpEF with CA and 12 healthy volunteers.

During a run-in phase up to 6 participants will be enrolled to standardise the trial procedures, especially mangafodipir-enhanced imaging.

The number and sequence of trial visits will be the same for participants of the run-in and the main phase.

All enrolled participants will undergo gadolinium-enhanced imaging at Visit 2. A gadolinium-based contrast agent (authorised AMP) will be injected i.v. and T1 mapping and Extracellular Volume (ECV) measurement will be done for approximately 60 minutes.

Mangafodipir-enhanced mapping will be done at Visit 3. After baseline T2 mapping, mangafodipir trisodium injection (IMP) will be administered i.v. and T1 mapping, Saturation Recovery T1 weighted imaging for measurement of the uptake rate, and T2 mapping, will be done for approximately 90 minutes.

Clinical safety data will be collected throughout the trial; the participants will be followed up by a phone call 24+6 hours after Visit 3 for evaluation of late-appearing AEs.

The analyses of the images will be done by an investigator of the study team, blinded to the clinical data.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have given their signed declaration of consent and data protection declaration.
2. Males and females (postmenopausal or surgically sterile females) aged ≥ 18 years and ≤ 90 years
3. HFpEF (= LVEF > 50%) with NYHA (New York Heart Association) class I, II and III and objective evidence of cardial structural and/or functional abnormalities consistent with the presence of left ventricular (LV) diastolic dysfunction/raised LV filling pressures, including raised natriuretic peptides.
4. Patients with HCM or CA (according to current guidelines)
5. Kidney functions eGFR (Estimated Glomerular Filtration Rate) > 30 mL/min/1.73 m2
6. Healthy volunteers (cohort specific criteria): adults with no known pre-existing medical conditions.

Exclusion Criteria:

1. Tachycardia (heart rate > 100, R-R interval < 600 ms)
2. NYHA IV
3. Previous coronary artery disease requiring intervention, including history of myocardial infarction including septal reduction therapies
4. Severely reduced renal function, defined as eGFR < 30 mL/min/1.73 m2
5. Severely reduced liver function (Child-Pugh class C), especially severe obstructive hepatobiliary disease
6. Phaeochromocytoma
7. Advanced cancer (with short/medium term prognosis)
8. History of chest radiation therapy
9. Diabetic patients
10. Severe valvular disease
11. Previous heart surgery
12. Left ventricular assist device (LVAD)
13. Severe pulmonary disease
14. Hypersensitivity to any medicinal products containing gadolinium
15. Hypersensitivity to the active substance of the IMP or to any of the excipients
16. Contraindications to MRI, including implanted cardiac devices/pacemakers
17. Participants not able to follow instructions necessary to conduct the MRI
18. Women of childbearing potential
19. Participation in other clinical studies with investigational drugs either concurrently or within the last 30 days
20. Previous participation in this clinical trial
21. History of ongoing drug abuse or alcoholism
22. Legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope, and possible impact of the trial
23. Investigator site staff and sponsor directly involved in the conduct of the study and their family members.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-11-29 (Actual); Study Completion 2025-11-29 (Actual)

PRIMARY OUTCOMES:
To quantify the manganese uptake rate after administration of mangafodipir trisodium in all segments of the left ventricular wall. | Images to be captured during the trial MRI examinations (up to 60 to 90 minutes after the drug administration); image evaluations shall be executed remotely.
  Determination of the manganese uptake rate.

SECONDARY OUTCOMES:
Efficacy: Comparison of manganese uptake rate constant in healthy volunteers, HFpEF with HCM or CA. | Images to be captured during the trial MRI examinations (up to 60 to 90 minutes after the drug administration); image evaluations shall be executed remotely.
  Difference in the uptake rate constant between healthy volunteers, HFpEF with HCM or CA.
To assess the safety of mangafodipir trisodium injection based on AEs. | From AMP administration at Visit 2 to the end of the Follow-up period (1 day after Vist 3).
  Frequency and severity of adverse events (AE).
To assess the safety of mangafodipir trisodium injection based on injection site AEs. | From AMP administration at Visit 2 to the end of the Follow-up period (1 day after Vist 3).
  Frequency of injection site AEs.
To assess the safety of mangafodipir trisodium injection based on vital signs. | From AMP administration at Visit 2 to the end of the Follow-up period (1 day after Vist 3).
  Significant changes in vital signs.
To assess the safety of mangafodipir trisodium injection based on ECG. | From AMP administration at Visit 2 to the end of the Follow-up period (1 day after Vist 3).
  Significant changes in ECG.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Department of Cardiology, Rikshospitalet Sognsvannsveien 20, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No